CLINICAL TRIAL: NCT00924495
Title: Regulatory Central Mechanisms in Chronic Nonspecific Low Back Pain With Lumbar Dysfunction
Brief Title: Study Comparing Cortical Function and Dysfunction Tests in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, olavi airaksinen, MD, PhD Ass Proff, Head of the Department of Rehabilitation, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KUH5960429
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Nonspecific Low Back Pain
Keywords: low back pain; motor control; cortical regulation; transcranial magnetic stimulation
MeSH Terms: conditions — Low Back Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Cortical function (Active Comparator): Activity/inhibition of the cortex
  Interventions: Device: transcranial magnetic stimulation
- Cortical regulation (Active Comparator)
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — rTMS therapy daily for two weeks, five times per week each lasting for half an hour

SUMMARY:
The purpose of this study is to explore the cortical regulation of the paraspinal muscles in chronic low back pain. These (possible) changes in regulatory mechanisms are being compared to other motor control tests in order to determine whether correlations are found. Furthermore the patients are being treated with repetitive transcranial magnetic stimulation (rTMS) and tested afterwards. The purpose is to find out if rTMS-therapy is capable of normalizing motor control deficits.

ELIGIBILITY:
Inclusion Criteria:

* chronic nonspecific low back pain for at least six months
* male gender
* age 25-50 yrs
* average pain during last week 4-8/10 by VAS
* Oswestry disability index 20-80 %

Exclusion Criteria:

* former spinal operations
* rheumatic disease, marked spondylolysis and -olisthesis, other diseases that markedly reduce physical or psychological performance, history of epilepsy, history of taking epileptic or strong opioid drugs

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Correlation between cortical activity and other motor control tests | day 1 and day 19

SECONDARY OUTCOMES:
The effect of rTMS-therapy for clinical outcome and motor control tests | day 19, 1 month, 2 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marja T Kilpiäinen, MD, Principal Investigator — Kuopio University Hospital; Markku Kankaanpää, MD,PhD, Study Director — Tampere University Hospital; Olavi Airaksinen, MD, PhD, Study Chair — Kuopio University Hospital; Timo Miettinen, MD,PhD, Study Chair — Kuopio University Hospital; Eeva Leino, MD,PhD, Study Chair — Tampere University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland